CLINICAL TRIAL: NCT06957236
Title: Surgical Site Infection Outcomes in Robotic Natural Orifice Colorectal Resection - The NICE Trial
Brief Title: Surgical Site Infection Outcomes in Natural Orifice Intracorporeal Anastomosis and Extraction (NICE) Procedure - The NICE Trial
Status: Enrolling by invitation | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Eric M. Haas, Chief of the Division of Colon & Rectal Surgery, The Methodist Hospital Research Institute
Other Study IDs: PRO00038141
Record Dates: First submitted 2025-04-04; First posted 2025-05-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Diverticulitis; Surgical Site Infection; Surgical Site Infections; Colorectal Surgery; Robotic Surgical Procedures; Clinical Trials; Diverticulitis, Colonic; Diverticulitis Colon; Diverticulitis; Perforation, Bowel
Keywords: Natural Orifice Specimen Extraction; Intracorporeal Anastomosis; Robotic Colorectal Surgery; Left Colectomy; Rectosigmoid Resection; Benign Colorectal Disease; Diverticulitis; Minimally Invasive Surgery; Surgical Site Infection; Surgical Outcomes; Robotic Surgery Outcomes
MeSH Terms: conditions — Diverticulitis; Surgical Wound Infection; Diverticulitis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NICE Procedure Cohort: This cohort includes patients undergoing elective left-sided colectomy or rectosigmoid resection for benign disease using the robotic Natural Orifice Intracorporeal Anastomosis and Extraction (NICE) procedure. The procedure involves robotic intracorporeal anastomosis and transrectal specimen extraction. No comparator or control group is used. Data collected will assess surgical site infection rates and recovery outcomes.

SUMMARY:
The goal of this observational study is to learn if a new surgical technique, called the NICE procedure, is as safe as standard methods for treating benign left-sided colon and rectal diseases in adults. The main question it aims to answer is:

Does the NICE procedure lead to similar or lower rates of surgical site infections (SSIs) within 30 days compared to traditional surgery?

Researchers will gather information from hospitals across the country to evaluate how well this procedure works when performed by experienced surgeons in everyday clinical settings.

Participants will:

Have surgery using the NICE procedure, which uses a robotic platform and removes the specimen through a natural opening (the rectum).

Be monitored for any infections or complications after surgery.

Complete surveys to track their recovery, bowel function, and quality of life for up to 6 months.

This study may help improve recovery, reduce pain, and lower infection risk in future colorectal surgeries.

DETAILED DESCRIPTION:
Background and Rationale The Natural Orifice Intracorporeal Anastomosis and Extraction (NICE) procedure represents an emerging innovation in minimally invasive colorectal surgery. It combines robotic intracorporeal anastomosis (ICA) with natural orifice specimen extraction (NOSE), typically transrectal, to avoid the need for an abdominal extraction incision. This approach may reduce surgical site trauma, postoperative pain, opioid use, and rates of incisional hernias.

Intracorporeal anastomosis has been widely studied in right-sided colectomies, with consistent evidence showing reduced surgical site infections (SSIs) and improved recovery. However, application to left-sided resections introduces unique challenges. The bacterial density in the left colon and rectum, combined with transrectal manipulation, may increase the risk of deep or organ-space SSIs. While early single-center experiences suggest the NICE procedure may be safe and effective, multicenter validation in a broader clinical setting is needed.

Study Objectives The primary objective of this study is to determine the 30-day incidence of surgical site infections (superficial, deep, and organ-space) in patients undergoing robotic left-sided colorectal resections using the NICE procedure. Secondary objectives include assessment of intraoperative technical performance, perioperative complications, postoperative recovery, and longer-term functional and quality of life outcomes.

Study Design This is a prospective, multicenter, observational cohort study enrolling patients undergoing elective robotic-assisted left colectomy or rectosigmoid resection for benign colorectal disease. All procedures will use the standardized NICE technique. Participating surgeons must have performed at least 20 prior NICE procedures. The study will run over a 24-month accrual period, with each patient followed for at least 6 months postoperatively.

Study Procedures Surgical intervention involves robotic left-sided resection with intracorporeal anastomosis and transrectal specimen extraction. All sites will follow a standardized Enhanced Recovery After Surgery (ERAS) protocol tailored to robotic colorectal surgery. Operative videos will be collected for quality control, ensuring adherence to the defined NICE procedural steps.

Postoperative follow-up includes in-person or remote assessments at 30 days, 3 months, and 12 months. Functional outcomes will be measured using validated questionnaires: Wexner score for fecal incontinence, LARS score for bowel dysfunction, and PROMS-10 for health-related quality of life.

Data Collection and Oversight Clinical data will be collected prospectively using REDCap, a secure, HIPAA-compliant electronic data capture system. All patient data will be pseudonymized. A centralized coordinating center will oversee data integrity, standardization, and site compliance. Surgical cases will be video recorded to ensure procedural fidelity.

Each site must consecutively enroll eligible patients and maintain compliance with protocol-defined ERAS standards. Surgeons will be credentialed based on review of unedited operative videos prior to participation.

Outcomes The primary outcome is the 30-day SSI rate, including superficial, deep, and organ-space infections. Secondary outcomes include intraoperative variables (e.g., operative time, blood loss, conversion rate), postoperative recovery (opioid use, length of stay, complications, readmissions, reinterventions), and long-term outcomes such as hernia formation and bowel function.

Patient-reported outcome measures will be collected preoperatively and at designated follow-up intervals. These include the Wexner score, LARS score, and PROMS-10, allowing for longitudinal evaluation of continence, function, and quality of life.

Sample Size and Statistical Considerations The study is powered to detect non-inferiority in SSI rates compared to conventional techniques. Assuming a historical SSI rate of 5% and a non-inferiority margin of 5%, a sample size of at least 224 patients provides 80% power with a 5% alpha. To accommodate multivariate modeling and variability across sites, the planned enrollment target is 300-400 patients.

Data will be analyzed using multilevel logistic regression to account for center and surgeon-level effects. Sensitivity analyses will be conducted to test robustness of findings. Descriptive and inferential analyses will be used to evaluate changes in quality of life and functional outcomes over time.

Significance This trial aims to provide high-quality evidence on the safety and performance of the NICE procedure for left-sided colorectal surgery. If non-inferiority is demonstrated, the findings may support broader adoption of this technique, with implications for faster recovery, reduced SSI risk, and improved patient experience. By incorporating video-based quality control and standardized ERAS pathways, the study ensures procedural consistency and real-world applicability of results.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis: Patients must be diagnosed with benign left-sided colon and rectosigmoid disease, including diverticulitis and benign colon neoplasia.

2. Age Requirement: Patients aged 18 years or older. 3. Cancer-Free: There must be no evidence of cancer or metastatic disease in the patients. This includes:

* Colonoscopy with no evidence of malignant lesion in the last 12 months
* CT scan with no concern for malignancy in the prior 6 months
* No other clinical concern for possible malignancy 4. Surgical Eligibility: Patients must be eligible to undergo robotic left colectomy with primary anastomosis without a planned diverting stoma.

  5. Informed Consent: Participants must be able to understand and willing to sign a written informed consent form.

  6. Treatment with NICE: Patients who undergo surgical treatment specifically with the NICE procedure.

  7. Surgeon Experience: The patients should be treated by surgeons who have performed at least 20 NICE procedures.

  8. General Practice Inclusion: Patients treated by surgeons who offer the NICE procedure as part of their general surgical practice and do not super-select patients for the procedure.

Exclusion Criteria

1. Urgent or emergent procedure
2. Patients diagnosed with cancer or metastatic disease are not eligible for the study. This includes:

   * Known genetic predisposition to colorectal cancer
   * First-degree family history of colorectal cancer
   * Any concern about colorectal cancer
3. Patients with an ongoing infection other than diverticulitis (e.g., pneumonia) or taking antibiotics unrelated to diverticulitis.
4. Patients with a history of pelvic radiation
5. Patients with prior anorectal surgery or prior colorectal surgery
6. Patients with fecal incontinence, outlet obstructive defecation, anismus, or levator spasm at baseline are excluded from the study
7. Any procedure in which a primary anastomosis is not feasible or diversion of the fecal stream is anticipated
8. Patients with a high ASA of 4 or more and clinical frailty score of 8 or more
9. Patients requiring preoperative nutritional support, such as total parenteral nutrition (TPN) or enteral feeding via percutaneous endoscopic gastrostomy (PEG) or nasogastric (NG) tube within 30 days prior to surgery
10. Systemic steroids used within the last 12 months or immunomodulators and biological agents used within the last 60 days prior to surgery will render the patient ineligible for the trial.

    * Preoperative antibiotics used within two weeks to treat diverticulitis are permitted.
    * Antibiotics used within 30 days before surgery for any condition other than treating an infection related to diverticulitis will render the patient ineligible for the trial.
11. Regional block anesthesia (e.g., epidural and spinal) is not permitted in this trial.
12. Chronic Opioid Use: Chronic use of opioids in the prior 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from multiple high-volume colorectal surgery centers across the United States that routinely perform robotic-assisted procedures. All participating sites follow a standardized Enhanced Recovery After Surgery (ERAS) protocol and are required to have surgeons experienced in the NICE procedure. The study population will consist of patients scheduled for elective robotic left-sided colectomy or rectosigmoid resection for benign disease, treated in real-world, non-super-selected surgical practice settings.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
30-Day Surgical Site Infection (SSI) Rate Following the NICE Procedure | 30 days post-surgery
  Measures the proportion of patients who develop surgical site infections (SSIs) categorized as superficial, deep, or organ-space within 30 days following robotic left-sided colectomy or rectosigmoid resection using the NICE procedure. Infections are classified per CDC definitions and assessed through clinical evaluation, medical records, and follow-up.

SECONDARY OUTCOMES:
Long-Term Outcomes: Hernia, Bowel Dysfunction, Fecal Incontinence | Up to 6 months post-surgery
  Monitors incidence of incisional hernia, long-term bowel dysfunction, and persistent fecal incontinence following the NICE procedure.
Stool Contamination Grade During NICE Procedure | During surgery
  Assesses the degree of fecal contamination encountered intraoperatively using a standardized grading scale.
  Scale Components and Interpretation:
  Degree of Contamination (Severity of contamination encountered):
  * 1 = Mild (Minimal stool, easily managed with minimal delay)
  * 2 = Moderate (Requires additional cleaning, minor to moderate delays)
  * 3 = Severe (Substantial contamination, extensive cleaning and procedural delay required) Higher scores indicate worse contamination.
  Quality of Contamination (Consistency of stool):
  * Liquid = Easily aspirated
  * Semi-formed = Partially cleared with aspiration
  * Solid = Requires transrectal/manual clearing
  Degree of Evacuation (Effectiveness of stool clearance):
  * Complete = All visible stool removed
  * Semi-complete = Minimal residual stool
  * Incomplete = Moderate residual stool
Estimated Intraoperative Blood Loss | During surgery
  Records the estimated blood loss in milliliters during the NICE procedure as documented by the surgical team.
Total Operative Time | During surgery
  Measures the total duration of the NICE procedure from skin incision to closure, reported in minutes.
Success Rate of Intracorporeal Anastomosis | During surgery
  Captures whether the intracorporeal anastomosis (ICA) was successfully completed as intended using the robotic platform.
Success Rate of Transrectal Specimen Extraction | During surgery
  Measures whether the surgical specimen was successfully extracted through the rectum without conversion to transabdominal extraction.
Incidence of Intraoperative Complications | During surgery
  Reports the occurrence of intraoperative complications such as rectal tear, sphincter injury, or conversion to open surgery.
Total Opioid Use Within 30 Days Post-Surgery | 30 days post-surgery
  Measures the cumulative opioid consumption during the first 30 days following surgery, expressed in morphine milligram equivalents (MME).
Length of Hospital Stay | 30 days post-surgery
  Measures the number of days from the date of surgery to the date of discharge, assessing early recovery and discharge readiness.
Overall Postoperative Complication Rate | 30 days post-surgery
  Proportion of patients who experience one or more postoperative complications, including minor and major events, within 30 days of surgery.
Reoperation or Re-intervention Rate | 30 days post-surgery
  Proportion of patients who require unplanned surgical reoperation or interventional procedures (e.g., drainage) within 30 days post-surgery.
Readmission Rate Within 30 Days | 30 days post-surgery
  Percentage of patients who are readmitted to any hospital for any cause within 30 days following the index surgery.
Postoperative Mortality Rate | 30 days post-surgery
  Percentage of patients who die from any cause within 30 days following the surgical procedure.
Use of Transrectal Wound Protector | During surgery
  Documents whether a wound protector was used during transrectal specimen extraction as part of the NICE procedure.
Type of Intracorporeal Anastomosis Staple Line | During surgery
  Classifies the anastomosis as either crossing or non-crossing staple line configuration.
Oversewing of Anastomosis | During surgery
  Indicates whether the anastomosis was reinforced with oversewing after stapling.
Performance of Mesenteric Shaving | During surgery
  Captures whether mesenteric shaving was performed on the specimen during the NICE procedure.
Change in Wexner Score for Fecal Incontinence | Baseline, 3 months, 12 months
  Evaluates changes in the Wexner score from baseline at 3 and 12 months to assess the severity and frequency of fecal incontinence following the NICE procedure. The Wexner score assesses the ability to control gas, liquid, and solid stool, the need for protective garments, and the impact on lifestyle.
  Scale Range: 0 (no incontinence) to 20 (complete incontinence); Higher scores indicate worse fecal incontinence.
Functional Outcomes: LARS Score | Baseline, 3 months, 12 months
  The Low Anterior Resection Syndrome (LARS) score assesses bowel dysfunction including incontinence, frequency, and urgency following low anterior resection. Evaluates changes over time.
  Scale Range: 0 to 42; Scores 0-20 indicate no LARS, 21-29 minor LARS, and 30-42 major LARS. Higher scores indicate worse bowel dysfunction.
Health-Related Quality of Life: PROMS-10 Score | Baseline, 3 months, 12 months
  PROMS-10 captures patient-reported physical, emotional, and social well-being using a 10-item questionnaire. Monitors change in health-related quality of life over time.
  Scale Range: 0 to 40; Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Haas, MD, Principal Investigator — The Methodist Hospital Research Institute; Muhammed Elhadi, MBBCh, Study Director — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the study team due to privacy concerns and the multicenter observational nature of the study. Although data are pseudonymized, the complexity and volume of surgical video and clinical data could still risk indirect identification. Data access is restricted to investigators approved by the study's steering committee to ensure confidentiality and ethical compliance.